CLINICAL TRIAL: NCT02958046
Title: Phase 4 Study, Assessing the Efficacy of Lansoprazole and Domperidone Combination on Intragastric and Intraesophageal Acidity
Brief Title: The Efficacy of Lansoprazole and Domperidone Combination on Intragastric and Intraesophageal Acidity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neu-01.13
Record Dates: First submitted 2015-09-01; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-10

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Lansoprazole; Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lansoprazole/Domperidone (Experimental): DUOLANS 30/30 mg SR tablet per oral, one tablet daily
  Interventions: Drug: Lansoprazole/Domperidone

INTERVENTIONS:
Drug: Lansoprazole/Domperidone — DUOLANS 30/30 mg SR tablet per oral, one tablet daily
  Other Names: Duolans

SUMMARY:
The purpose of this study is to investigate the efficacy of lansoprazole combination with domperidone on intragastric acidity and intraesophageal acidity, GERD symptoms, impedance kinetics, gastric emptying in patients with gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
Objectives of the trial to assess the efficacy of lansoprazole in combination with domperidone on gastric acidity, intraesophageal acidity, GERD symptoms, impedance kinetics and gastric emptying in patients with GERD.

24 hour pH measurement and gastric emptying test will be done at screening visit and after 7 days of drug treatment. Twelve patients will take one tablet for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GERD with symptoms (i.e. regurgitation, pyrosis) during last one year with at least 1 or more episodes a week
* Age ≥ 18 years and <65 years
* Helicobacter pylori (an infection) negative
* Have a body mass index (BMI) between 18 and 33 kg/m²
* pH>4 gastric exposure <25% on a 24-hour dual pH channel monitoring study performed prior to screening (normal intragastric pH +2SD)
* Pathologic intraesophageal acidity exposure (DeMeester score >14.75 and/or >4% of pH<4 (at least 21 hours measured)

Exclusion Criteria:

* Have food existence at stomach during upper GIS endoscopy, Barrett's stricture, GIS bleeding, malignite, and all type of GIS pathology to affects the study
* Have allergy to the study drug or any of the excipients of the formulation
* Must use of pain relieving medications (NSAIDs) during study, (paracetamol not excess of 2 gram/day can be used)
* Use of any concomitant therapy which are drug affects the motility of GIS and acid secretion
* Use of prostaglandin analogs and sucralfate
* Have taken PPIs or H2-blockers within 7 days and prokinetic drugs within 3 days before entering the study
* History of surgery of cholecystectomy
* Abusing drugs or alcohol
* Have a major psychiatric disease
* Use of antidepressant (patient with minor depression or under controlled with drug can be included)
* Have suppressed immune system or taken a immunosupressive treatment, including cortisone.
* Have malabsorption, gastric outlet obstruction that affects the absorption of drug
* Must use of drug ketoconazole, iron salts, digoxin, ampicilin esters , anticoagulants, antineoplastic agents
* Women who are pregnant or of childbearing
* Have gastroparesis
* Current or a history of cancer, with the exception of fully excised skin carcinoma (Malign Melanoma will be excluded).
* Have severe concomitant disease (i.e. uncontrolled or insuline dependent diabetes mellitus, symptomatic bladder stone (patients have asemptomatic, not undergone colesistit, stone <3cm and polib <1cm can be included), active or unhealed gastric or duodenum ulcer, Zollinger Ellison syndrome, primary esophageal motility disorder, pancreatitis, inflammatory bowel disease, chronic hepatic disease, severe lung disease, uncontrolled kidney failure, cardiac failure, cerebrovascular disease, epilepsy) which affects the conduct and result of study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The percentage time of 24-hour intragastric pH >4 compared to baseline | 7 days
The AUC of 24-hour intragastric pH >4 compared to baseline | 7 days

SECONDARY OUTCOMES:
The significant increase in total measurements of median pH | 7 days
The significant increase in nocturnal measurements of median pH | 7 days
The decrease in reflux symptom index calculated by weekly regurgitation numbers | 7 days
The decrease in reflux symptom index calculated by weekly pyrosis numbers | 7 days
The percentage time of 24-hour intragastric pH >2 compared to baseline | 7 days
The percentage time of 24-hour intragastric pH >6 compared to baseline | 7 days
The AUC of 24-hour intragastric pH >2 compared to baseline | 7 days
The AUC of 24-hour intragastric pH >6 compared to baseline | 7 days
The percentage time of 24-hour total intragastric pH >4 compared to baseline | 7 days
The AUC of 24-hour total intragastric pH >4 compared to baseline | 7 days
The evaluation of gastric emptying by octanoic acid breath test compared to baseline | 7 days
The evaluation of safety of study drug (Number of Participants with Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment) | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Neutec Ar-Ge San ve Tic A.S, Study Director — Neutec Ar-Ge Clinical Trial
Locations (1):
- Department Of Gastroenterology, Faculty Of Medicine, Ege University, Izmir, Turkey, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided